CLINICAL TRIAL: NCT02407067
Title: A Comparison of Voice Amplifiers and Personal Communication Systems in Individuals With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Scott Adams, Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 106169
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Parkinson's Disease; Dysarthria
MeSH Terms: conditions — Parkinson Disease; Dysarthria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Voice Amplifier (Active Comparator): Participant will be fit with a voice amplifier (ChatterVox) and it will be used during speech testing and during regular conversations over a one week period.
  Interventions: Device: ChatterVox
- Personal Communication System (Experimental): Participant will be fit with a personal communication system (Easy Listener FM system) and it will be used during speech testing and during regular conversations over a one week period.
  Interventions: Device: Easy Listener FM system (Phonic Ear Corp.)

INTERVENTIONS:
Device: ChatterVox — A voice amplifier will be attached to the participant and used for the treatment of low speech intensity (hypophonia) and reduced speech intelligibility in Parkinson's disease.
  Other Names: Voice Amplifier
  Arms: Voice Amplifier
Device: Easy Listener FM system (Phonic Ear Corp.) — A personal communication (FM) system will be attached to the participant and used for the treatment of low speech intensity (hypophonia) and reduced speech intelligibility in Parkinson's disease.
  Personal Communication System
  Arms: Personal Communication System

SUMMARY:
This study will compare two types of assistive devices for communication (a voice amplifier and a personal communication system) in individuals with a speech disorder related to Parkinson's disease. The performance of these two devices will be examined with measures of speech intelligibility and patient questionnaires and rating scales.

DETAILED DESCRIPTION:
The proposed study will involve a comparison of 2 types of communication devices that are approved for use in individuals with communication disorders. One of the devices, the voice amplifier, is frequently prescribed for individuals with Parkinson's disease and should be considered as part of the standard care for the symptom of low speech intensity in this disorder. The other device is frequently prescribed for individuals with hearing impairment (unrelated to Parkinson's disease) but is not considered to be part of the standard of care for individuals with Parkinson's disease. This clinical study will use a crossover design in which the participants will receive both devices, one after the other, and the order will be randomized across the individuals. There is no control group or placebo.

This study will include three groups of participants: 1) a PD participant group (n=20), 2) a communication partner (CP) group (n=20), and 3) a naïve listener group (n=10). The PD participant group will be comprised of individuals who have mild to moderate signs and symptoms of idiopathic PD and hypophonia as confirmed by a neurologist. For all individuals with PD, the speech testing will occur approximately one hour after taking their antiparkinsonian medication according to their regular medication schedule. The communication partner group will consist of individuals who regularly converse with the PD participant (i.e. spouse or primary caregiver). The naive listener group will consist of students from Western University. The participants with PD will wear a head-set microphone (AKG c520). The speech intensity of the participants with PD will be calibrated with a sound level meter (Luton SL-4001) placed 15cm from the mouth while the participant produces a steady 70dB A prolonged "ah" for about 2 seconds. Two additional tripod-mounted microphones (Shure SM48) will be placed 2 meters and 4 meters from the PD participant. The communication partner participants will be seated approximately 30cm from these two microphones during the 2 and 4 meter interlocutor distance conditions. The output from the 3 microphones will be connected to preamplifiers and a digitizing unit (M-Audio MobilePre) attached via a USB connection to a PC computer running Praat recording and analysis software (Boersma & Weenink, 2013). An additional, fourth input line will be attached to the digitizing unit from the output of the personal communication system when this device is being used in the study. All four audio signals will be digitized at 44.1 kHz and 16 bits and stored as uncompressed .wav audio files. The voice amplifier and personal communication system will be evaluated in random order across the participants. The voice amplifier will be a ChatterVox. This amplifier includes a headset microphone wired to a speaker/amplifier unit that is worn on a waist belt. The ChatterVox was selected because it is a typical type of voice amplifier that is frequently recommended and prescribed to individuals with PD in Ontario. Despite the paucity of published voice amplifier studies of PD, the ChatterVox has been used in several published studies of non-neurological voice disorders such as studies of elementary school teachers with occupational-related voice problems (McCormick & Roy, 2002; Roy et al. 2003). In addition, a recent MSc thesis conducted at Western University by Monika Andreetta (supervised by Professor Scott Adams) found that the ChatterVox was one of the best performing and preferred devices in participants with PD when it was compared to 6 other voice amplifiers. The personal communication system that will be evaluated is the Easy Listener FM system (Phonic Ear Corp.). This system includes a light-weight, pocket-sized (2.5 x 9.4 x 5.6 cm; 80 grams) transmitter unit with a head-set microphone and a nearly identical, pocket-sized receiver unit with a set of small headphones. These units can be carried in a breast-pocket or attached to a waist-belt with a clip. The transmitter and receiver units are wireless and communicate via an FM signal. The communication range of the units is approximately 30 meters. The PD participant will wear the transmitter/microphone unit and the communication partner (CP) participant will wear the receiver/headphone unit. While there are several personal communication systems that are available, the Easy Listener personal communication system has been frequently prescribed and has been used in several previous studies of individuals with hearing impairment (Schafer & Thibodeau, 2004). During some of the experimental conditions the PD and CP participants will be presented with 65dB A of multi-talker noise (using a standard Audiotec Corp. Recording of 4-talker noise). The noise will be presented from a computer via an audio amplifier and loudspeaker placed at 2 meters from the participants. A sound level meter will be used to calibrate the noise level from the loudspeaker. Procedures: Speech Tasks: Once one of the two devices has been attached to the participant(s), the PD participant will be given a list of 6 sentences that were randomly generated from the Sentence Intelligibility Test software. The PD participant will read aloud each sentence and then pause while the communication partner (CP) participant attempts to repeat aloud the sentence. The SIT provides intelligibility measures, which are commonly used to document effectiveness in intervention programs or outcome studies (Beukelman et al., 2007). Furthermore, most of the supportive research for the SIT was completed with dysarthric speakers (Beukelman et al., 2007). After the list of 6 sentences are completed the PD participant will be given several pictures of people engaged in various activities (i.e. fishing, playing baseball, doing dishes, etc.) and the PD participant will make statements that describe the pictures while the CP participant repeats aloud each of these statements. This will continue until 6 statements (minimum of 5 words each) have been produced/repeated. Speech Conditions: The speech tasks will be repeated with no device and while using each of the two devices (ChatterVox voice amplifier and Easy Listener personal communication system) in two noise conditions (none and 65dB multi-talker noise) and two interlocutor distances (2 and 4 meters). These conditions will be randomized. Rating Scale Procedures: Immediately following the speech tasks the PD and CP participants will be asked to rate their experience with the devices using visual analogue scales related to the following five parameters: 1. Physical comfort: uncomfortable versus comfortable 2. Visual presentation: unacceptable versus acceptable 3. Sound quality: poor sound quality versus good sound quality 4. Amplification power: poor amplification versus good amplification 5. Overall preference: low preference versus high preference The PD and CP participants will use the five visual analogue scales to provide separate ratings for each of the two devices. Following the completion of the rating scales the participants will be encouraged to provide additional feedback about their impressions of the 2 devices. One Week Trial Periods: After the completion of the lab-based speech and rating scale procedures the PD and CP participants will be given instructions on the care and use of one of the two devices (i.e. recharging, cleaning, volume adjustments, attachment, positioning, etc.) and then take the device home for a one week trial period. The participants will be asked to use the device as often as they desire but to use the device at least 3 times for a periods of at least one hour over the course of the week. The participants will be given a Device Use Diary to write down the dates, times, volume settings and contexts that they used the devices. The participants will return after one week and complete questionnaires and rating scales related to their experience and evaluation of the device. These will include the following: 1. Visual analogue scales related to physical comfort, visual presentation, sound quality, amplification power, and overall preference. 2. Speech Amplification Satisfaction Scale 3. Quebec User Evaluation of Satisfaction with Assistive Technology Scale 4. Psychosocial Impact of Assistive Devices Scale (PIADS). Following the completion of these questionnaires and ratings scales, the participants will be given instructions on the use and care of the second device and then take the device home for another one week trial period. The participants will be asked to use the device as often as they desire but to use the device at least 3 times for a periods of at least one hour over the course of the week. The participants will be given a Device Use Diary to write down the dates, times, volume settings and contexts that they used the devices. The participants will return after one week and again complete the previously described questionnaires and rating scales related to their experience and evaluation of the device.

Listening Tasks: Listener participants will listen to pre-recorded speech samples obtained from the tripod-mounted microphones. Speech samples will be played in a randomized order. Listeners will not be present at the time speech samples are recorded, and they will be blinded to all information about the speakers and to the contents of the sentences from both the SIT and picture description tasks prior to hearing them. Listeners will be seated at a comfortable distance from a loudspeaker, which will be fixed at a comfortable predetermined volume, and they will be asked to transcribe the data orthographically on prepared forms that will be numbered to match the presentation order of the stimuli. The SIT software will compute an intelligibility score by comparing transcribed words and sentences to the stimuli on the master lists. For the picture description task, sentences will be transcribed independently by the assessor and then compared to the listeners' transcriptions to determine the intelligibility score.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Parkinson's disease by a neurologist at least 6 months prior to testing • Exhibit mild to moderate signs and symptoms of Parkinson's disease and hypophonia (reduced speech intensity) • Stabilized on antiparkinsonian medication

Exclusion Criteria:

* Exhibit severe signs and symptoms of Parkinson's disease • History of stroke or an additional neurological or motor control disorder • History of speech impairment that is unrelated to Parkinson's disease

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Speech Intelligibility Score | up to 5 min
  The Sentence Intelligibility Test will be used to obtain speech intelligibility scores (%) while participants are speaking and using the two communication devices during quiet and 65 decibels of multi-talker background noise. Speech intelligibility scores will be obtained from communication partners who will provide live repetitions of the participant's spoken sentences and from listener transcriptions of the participant's audio recorded spoken sentences.
Device Performance Rating Score | 30 minutes and 7 days
  Visual analogue scales related to physical comfort, visual presentation, sound quality, amplification power, and overall preference will be used by the participant with Parkinson's disease and the associated communication partner to evaluate the devices following the initial 30 minutes of use (treatment) and following 7 days of use (treatment).
Device Satisfaction Rating Score | 7 days
  The Speech Amplification Satisfaction Scale and the Quebec User Evaluation of Satisfaction with Assistive Technology Scale will be used by the participant with Parkinson's disease and the associated communication partner to evaluate the devices following 7 days of use (treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Scott G Adams, PhD, Principal Investigator — Western University, Canada

IPD SHARING:
Plan to Share IPD: No